CLINICAL TRIAL: NCT00812734
Title: Etude épidémiologique Multicentrique Des Douleurs Neuropathiques Post-opératoires
Brief Title: Epidemiologic Multicentre Study of Neuropathic Post-surgical Pain
Acronym: EDONIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CHU-0044
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2013-04

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic pain; chronic pain; postoperative; surgery; anesthesiology; Scheduled surgery
MeSH Terms: conditions — Neuralgia; Chronic Pain | interventions — Blood Specimen Collection; Genome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- surgery
  Interventions: Procedure: Blood sampling for genomics; harvesting of a sample of intercostal muscle for proteomics (thoracotomies only)

INTERVENTIONS:
Procedure: Blood sampling for genomics; harvesting of a sample of intercostal muscle for proteomics (thoracotomies only) — Blood sampling for genomics; harvesting of a sample of intercostal muscle for proteomics (thoracotomies only)

SUMMARY:
This cohort study aims to know the prevalence at 3 and 6 months after surgery, of persistent pain, as well as to describe the neuropathic features of this pain. It includes more than 3000 patients scheduled for different types of surgery, some of them already known to induce persistent pain, some being frequent procedures with no additional data. Clinical and genetical risk factors will be searched.

DETAILED DESCRIPTION:
Neuropathic post-surgical pain (NPSP) motivates the consultation of the French Centres for Evaluation and Treatment of Pain in 20 to 35% of the cases. The following table shows the available data of literature about chronic post-surgical pain:

Surgery Prevalence of chronic pain (%) Neuropathic symptoms Mastectomy 22 to 49 Yes Inguinal hernia repair 30 to 63 Yes Sternotomy 28 to 40 Unknown Saphenectomy 5 to 7 Yes Mandibular osteotomy Unknown Yes Cholecystectomy 3 to 20 Unknown Caesarean section 6 Unknown Thoracotomy 50 to 75 Yes Knee arthroscopy Unknown Unknown Rectal amputation 12 to 18 Unknown Limb amputation 60 Yes Endodontic treatment 5 to 13 Unknown

In most of these cases, the mechanism of pain is highly suspected as neuropathic, although the location of the nerve(s) concerned is unclear. However, the clinical features of the pain are often poorly described. In other types of surgery (such as caesarean section or cholecystectomy), the report of chronic pain may be related to the high frequency of these procedures.

The initiation of NPSP can be identified on a time scale (i.e. day of surgery), and can be prospectively expected. This leads to possibility of (i) a better understanding of the evolution of neuropathy following time and (ii) a study of putative preventive (peritraumatic) treatments. Thus, NPSP appears as strongly different from other chronic pain syndromes (such as diabetes mellitus, chemotherapy for cancer or even post-traumatic) for which the time course, mechanisms and psychic interactions are more complex.

We suspect that overall prevalence of NPSP may have been underestimated, as (i) the delay of onset of pain may be in a range between some days to several months, (ii) there is not always a systematic follow-up after most of the surgical procedures, and patients may stay out of the medical network and (iii) the benefit provided by the surgical procedure may lead to patient not to complain from a somewhat "necessary" complication.

No large epidemiologic study has been performed concerning neuropathic post-surgical pain at this date. The principal aim of this study is to know the exact prevalence of NPSP, 3 and 6 months after the date of surgery. Only nine surgical procedures have been considered for the study, according to the previous data of literature and/or the high frequency of practice. This is a prospective open epidemiologic study, performed in nine French university general hospitals, three anti-cancer university hospitals and many other general hospitals. The secondary endpoints are (i) to find a relationship (by multivariate analysis) between NPSP and a large number of clinical/biological items (quality of life, habits, treatments, drug abuse, psychic/mental state, genome…) collected preoperatively, (ii) to validate a self-completed version of a questionnaire already validated for discriminating the neuropathic feature of chronic pain (DN4), and (iii) to assess the availability of the existing medical networks for the care of NPSP.

Patients (age > 18) scheduled for one of the nine types of surgery will be recruited. The number of patients (following table) to be recruited has been calculated on the basis of the reported prevalence of pain in literature (set to 20% if no data were available), with a risk set to 5%, a precision measure set to 5% and a prediction of 20% of lost patients during the study.

Type of surgery Number requested Caesarean section 103 Inguinal hernia repair (under laparoscopy) 389 Inguinal hernia repair (without mesh) 389 Inguinal hernia repair (with mesh) 389 Mastectomy (simple without axillary node dissection) 454 Cholecystectomy (under laparoscopy) 297 Saphenectomy (excluding harvesting for coronary bypass) 167 Sternotomy 374 Thoracotomy 463 Knee arthroscopy 297 Total 3322

The anaesthetist in charge of the patient during the pre-anaesthetic visit will complete the data sheet concerning the preoperative status of the patient. He will proceed to the inclusion and provide the data concerning the anaesthetic and analgesic protocol that have been followed. The inclusion will be registered by the local coordinating assistant, who will (i) send to the patient self-questionnaires 3 and 6 months after the date of surgery (about pain, neuropathic symptoms and the resulting quality of life) and (ii) transfer the information to the national coordinating centre (Centre for Clinical Investigations of Clermont-Ferrand). A permanent monitoring of inclusions and follow-up will be performed at both local and national levels. This will help to organise the rhythm and the location of inclusions at any time of the study.

If a case of chronic pain is identified, the willing patient will be sent to the closest Centre for Evaluation and Treatment of Pain, in which the diagnosis will be completed and a treatment initiated if required. For the validation of the self-completed version of the DN4 questionnaire, data from painless, painful neuropathic, and painful non-neuropathic patients, will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to the study
* Scheduled for one of the following surgeries :

  * caesarean section
  * inguinal hernia repair
  * mastectomy
  * cholecystectomy under laparoscopy
  * saphenectomy (excluding harvesting for coronary bypass)
  * sternotomy
  * thoracotomy
  * knee arthroscopy
* Major over 18 years

Exclusion Criteria:

* Emergency
* Inability to fill questionnaires
* Unreachable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Definied population
Sampling Method: Probability Sample
Enrollment: 3322 (Actual)
Dates: Start 2006-04; Primary Completion 2010-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Rate of persistent pain at 3 and 6 months after surgery | at 3 and 6 months after surgery

SECONDARY OUTCOMES:
Rate of persistent neuropathic pain at 3 and 6 months after surgery. Identification of risk factors collected before surgery. Links with genome. | at 3 and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christian Dualé, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Niccolai P, Ouchchane L, Libier M, Beouche F, Belon M, Vedrinne JM, El Drayi B, Vallet L, Ruiz F, Biermann C, Duchene P, Chirat C, Soule-Sonneville S, Duale C, Dubray C, Schoeffler P. Persistent neuropathic pain after inguinal herniorrhaphy depending on the procedure (open mesh v. laparoscopy): a propensity-matched analysis. Can J Surg. 2015 Apr;58(2):114-20. doi: 10.1503/cjs.008314. PMID 25799247
- [Derived] Blanc P, Genin E, Jesson B, Dubray C, Duale C; EDONIS-gene Investigating group. Genetics and postsurgical neuropathic pain: An ancillary study of a multicentre survey. Eur J Anaesthesiol. 2019 May;36(5):342-350. doi: 10.1097/EJA.0000000000000986. PMID 30882400
- [Derived] Richez B, Ouchchane L, Guttmann A, Mirault F, Bonnin M, Noudem Y, Cognet V, Dalmas AF, Brisebrat L, Andant N, Soule-Sonneville S, Dubray C, Duale C, Schoeffler P. The Role of Psychological Factors in Persistent Pain After Cesarean Delivery. J Pain. 2015 Nov;16(11):1136-46. doi: 10.1016/j.jpain.2015.08.001. Epub 2015 Aug 20. PMID 26299436
- [Derived] Lefebvre-Kuntz D, Duale C, Albi-Feldzer A, Nougarede B, Falewee MN, Ouchchane L, Soule-Sonneville S, Bonneau J, Dubray C, Schoeffler P. General anaesthetic agents do not influence persistent pain after breast cancer surgery: A prospective nationwide cohort study. Eur J Anaesthesiol. 2015 Oct;32(10):697-704. doi: 10.1097/EJA.0000000000000215. PMID 26053994
- [Derived] Duale C, Ouchchane L, Schoeffler P; EDONIS Investigating Group; Dubray C. Neuropathic aspects of persistent postsurgical pain: a French multicenter survey with a 6-month prospective follow-up. J Pain. 2014 Jan;15(1):24.e1-24.e20. doi: 10.1016/j.jpain.2013.08.014. Epub 2013 Oct 25. PMID 24373573